CLINICAL TRIAL: NCT00813865
Title: An Open-Label, Multicenter, Long-Term Extension Study To Assess The Safety, Efficacy, And Pharmacodynamics Of AT2101 In Adult Patients With Type 1 Gaucher Disease
Brief Title: A Long-Term Extension Study of AT2101 (Afegostat Tartrate) in Type 1 Gaucher Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GAU-CL-202X
Record Dates: First submitted 2008-12-22; First posted 2008-12-23 (Estimated); Results first posted 2018-08-15 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-07

CONDITIONS: Gaucher Disease; Type 1 Gaucher Disease; Gaucher Disease, Type 1
Keywords: Amicus Therapeutics; AT2101; afegostat tartrate; isofagomine tartrate
MeSH Terms: conditions — Gaucher Disease | interventions — AT2101

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Afegostat Tartrate Treatment Regimen 1 (Experimental): Afegostat tartrate was administered orally at a dose of 225 mg QD for 3 or 7 consecutive days followed by no study medication for 4 or 7 consecutive days (consecutive 3-days-on/4-days-off or 7-days-on/7-days-off, respectively). Amendment 2 added a MWF 3-days-on/4-days-off regimen. After Amendment 2 was implemented, all participants were assigned to one of the two 3-days-on/4-days-off regimens. Amendment 4 removed the consecutive 3-days-on/4-days-off regimen, and all participants were assigned to the MWF 3-days-on/4-days-off regimen. Participants were to receive afegostat tartrate for 30 months and be followed for 6 months after EOT.
  Interventions: Drug: afegostat tartrate

INTERVENTIONS:
Drug: afegostat tartrate
  Other Names: AT2101; isofagomine tartrate

SUMMARY:
This study evaluated the long-term safety and efficacy of afegostat tartrate in participants with Gaucher disease who were enrolled in a previous Phase 2 study of afegostat tartrate.

DETAILED DESCRIPTION:
This was an open-label, long-term extension study of afegostat tartrate in participants with type 1 Gaucher disease who successfully completed Study GAU-CL-202 (NCT00446550). Participants could enter the study immediately upon completion of participation in the lead-in study GAU-CL-202, or at any later time point. Participants received 225 milligram (mg) afegostat tartrate, administered orally for 30 months, and remained in 1 of the 2 randomized treatment regimens of Study GAU-CL-202: afegostat tartrate once daily (QD) for 3 consecutive days, then no afegostat tartrate for 4 consecutive days (consecutive 3-days-on/4-days-off) or QD for 7 consecutive days, then no afegostat tartrate for 7 days (consecutive 7-days-on/7-days-off). Amendment 2 removed the 7-days-on/7-days-off regimen and added an alternative 3-days-on/4-days-off regimen: afegostat tartrate QD on Monday, Wednesday, and Friday, then no afegostat tartrate on Tuesday, Thursday, Saturday, and Sunday (MWF 3-days-on/4-days-off). Once Amendment 2 was implemented at a site, participants assigned to the 7-days-on/7-days-off regimen switched to a 3-days-on/4-days-off regimen; those on the original 3-days-on/4-days-off regimen could switch to the MWF 3-days-on/4-days-off regimen. Amendment 4 removed the original 3-days-on/4-days-off regimen and any participants still on that regimen switched to the MWF 3-days-on/4-days-off regimen. Study visits occurred every 3 months for 30 months. Participants were contacted approximately 1, 3, and 6 months after the end of treatment (EOT) or early termination for follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants, 18 years of age or older
* Completed study GAU-CL-202 with no significant protocol violations or safety concerns
* Clinically stable
* Had not received enzyme replacement therapy (ERT) or substrate reduction therapy (SRT) in the past 12 months and was willing not to initiate ERT or SRT during study participation
* Agreed to practice an acceptable method of contraception
* Provided written informed consent to participate in the study

Exclusion Criteria:

* During the screening period, had any clinically significant findings which would compromise the safety of the participant, or preclude the participant from completing the study as deemed by the investigator
* Had a clinically significant disease, severe complications from Gaucher disease, or serious intercurrent illness that may preclude participation in the study, in the opinion of the Investigator
* Had a history of allergy or sensitivity to the study drug or any excipients, including any prior serious allergic reaction to iminosugars (for example, miglustat)
* Had a pacemaker or other contraindication for magnetic resonance imaging scanning
* Was pregnant or breast-feeding
* Had current gastrointestinal, liver, or kidney disease, sequelae of these diseases, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs
* Participant was otherwise unsuitable for the study in the opinion of the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-05-11 (Actual); Primary Completion 2012-05-01 (Actual); Study Completion 2012-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Amicus Therapeutics, Inc.
Locations (4):
- United States (3):
  - Coral Springs, Florida
  - Decatur, Georgia
  - Boston, Massachusetts
- London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were screened for evaluation of eligibility to participate in the study. Eight participants received at least 1 dose of study drug.
Groups:
- Afegostat Tartrate: Afegostat tartrate was administered orally at a dose of 225 milligram (mg) once daily (QD) on Monday, Wednesday, and Friday, with no study medication on Tuesday, Thursday, Saturday, and Sunday (MWF 3-days-on/4-days-off). Participants were to receive afegostat tartrate for 30 months and be followed for 6 months after the end of treatment (EOT).
Period: Overall Study
Arm/Group | Afegostat Tartrate
Started | 8
Safety Population (All participants who received at least 1 dose of study drug) | 8
Pharmacodynamic (PD) Population (Participants in the Safety Population with a baseline and at least 1 post-baseline PD measurement.) | 8
Completed | 1
Not Completed | 7
Not completed — Failure to Respond | 3
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- Afegostat Tartrate: Afegostat tartrate was administered orally at a dose of 225 mg QD MWF 3-days-on/4-days-off. Participants were to receive afegostat tartrate for 30 months and be followed for 6 months after EOT.
Arm/Group | Afegostat Tartrate
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (20.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Number Of Participants Who Experienced Severe Treatment-emergent Adverse Events (TEAEs)
Description: A TEAE was defined as any adverse event (AE) with start date on or after administration of study drug or pre-existing conditions that worsened on or after the start of the first study drug administration (on Day 1). A severe AE defined as an AE that was incapacitating and required medical intervention. The number of participants who experienced 1 or more severe TEAEs after dosing on Day 1 through the end of follow-up is presented. A summary of serious and all other non-serious AEs regardless of causality is located in the Reported Adverse Events module.
Time Frame: Day 1 (after dosing) through end of follow-up (6 months after EOT)
Population: Safety Population: all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Afegostat Tartrate
Number analyzed (Participants) | 8
Participants | 0

2. Secondary Outcome: Change From Baseline To EOT In Volume Of Spleen As Assessed By Magnetic Resonance Imaging (MRI)
Description: Standard MRI procedures were used to measure the volume of the spleen. The baseline value was defined as the value recorded on Days 1 to 3 of the study (certain values could have been carried over from the last assessment in the lead-in study, GAU-CL-202). A negative change from Baseline indicates that spleen volume decreased.
Time Frame: Baseline, Month 30
Population: PD Population: all participants in the Safety Population who had a baseline and at least 1 post-baseline PD measurement. Seven of 8 participants did not complete the study and did not contribute data to this endpoint.
Measure: Number; unit: cubic centimeters (cm^3)
Arm/Group | Afegostat Tartrate
Number analyzed (Participants) | 1
cubic centimeters (cm^3) | -138

3. Secondary Outcome: Change From Baseline To EOT In Volume Of Liver As Assessed By MRI
Description: Standard MRI procedures were used to measure the volume of the liver. The baseline value was defined as the value recorded on Days 1 to 3 of the study (certain values could have been carried over from the last assessment in the lead-in study, GAU-CL-202). A negative change from Baseline indicates that liver volume decreased.
Time Frame: Baseline, Month 30
Population: as for outcome 2
Measure: Number; unit: cm^3
Arm/Group | Afegostat Tartrate
Number analyzed (Participants) | 1
cm^3 | 57

ADVERSE EVENTS:
Time Frame: Day 1 (after dosing) through end of follow-up (6 months after EOT)
Arm/Group | Afegostat Tartrate
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 6/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afegostat Tartrate (N=8)
Splenomegaly (Blood and lymphatic system disorders) | 2
Splenic infarction (Blood and lymphatic system disorders) | 1
Blepharitis (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 1
Lacrimation increased (Eye disorders) | 1
Macular scar (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 2
Gait disturbance (General disorders) | 1
Hepatomegaly (Hepatobiliary disorders) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Muscle strain (Injury, poisoning and procedural complications) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
Due to the early withdrawal of 7 of the 8 study participants, there were no comparative data. Accordingly, no definitive conclusions regarding afegostat tartrate safety, efficacy, or pharmacodynamic effects can be made based on this information.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator can publish only the results from this trial, provided they supply the sponsor (or authorized entity) a copy of any proposed publication for review prior to submission for publication. If requested and prior to publication, the investigator will remove information deemed confidential or proprietary by the sponsor and will withhold publication for an additional period of time to allow the sponsor to take appropriate measures to establish and preserve its proprietary rights.